CLINICAL TRIAL: NCT00511017
Title: A Phase I Study of Doxercalciferol in Recurrent Pediatric Solid Tumors
Brief Title: Doxercalciferol in Recurrent Pediatric Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0423
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Doxercalciferol; Pediatric Cancer; Recurrent Pediatric Solid Tumors; Calcium; Vitamin D
MeSH Terms: conditions — Neoplasms | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxercalciferol (Experimental)
  Interventions: Drug: Doxercalciferol

INTERVENTIONS:
Drug: Doxercalciferol — .05 mcg/kg by mouth daily x 28 Days

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of doxercalciferol that can be given to pediatric patients with relapsed solid tumors. The safety of this drug will also be studied. Another goal is to measure the effect of the study drug on the blood levels of calcium and vitamin D.

DETAILED DESCRIPTION:
The Study Drug:

Doxercalciferol is designed to "copy the actions" of Vitamin D without causing blood levels of calcium to be too high.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will begin receiving doxercalciferol. The dose you will receive will be based on how many participants have been enrolled before you, and on the safety data that is available. You will remain on the same dose level throughout this study. There will be up to 9 participants enrolled in each group of the same dose. The first group of participants enrolled on this study will be given small doses of doxercalciferol. If no intolerable side effects are experienced, the next group of participants will be enrolled at a higher dose level. This process will continue until researchers find the highest tolerable dose of doxercalciferol, among the 5 dose levels being tested, that can be given without intolerable side effects occurring.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin the first "cycle" of the study drug. Each cycle of chemotherapy will last 28 days.

Doxercalciferol will be taken by mouth every day for 28 days.

Study Visits:

Every week during Cycle 1, you will have a physical exam, and urine will be collected for routine tests.

Two (2) times every week while you are on study, blood (about 2 teaspoons) will be drawn for routine tests.

During Cycles 2 and beyond, you will have the following tests and procedures performed:

* Urine will be collected for routine tests.
* ECG and ECHO will be repeated again only if your doctor feels it is necessary.
* You may also have a computed tomography (CT) scan and/or magnetic resonance imaging (MRI) to check the status of the disease.

Length of Study:

You may remain on this study for up to 12 cycles.You will be taken off this study if the disease gets worse or intolerable side effects occur. The study doctor may stop you from taking part in this study at any time if he/she believes it is in your best interest or if you do not follow the study rules.

You can stop participating in this study at any time. Tell the study doctor if you are thinking about leaving the study so that any risks can be reviewed by your study doctor and so that follow-up care and testing can be discussed. The study doctor will tell you how to stop safely.

End-of-Study Visit:

Once you are off-study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed.

* You will have a physical exam.
* Blood (around 2 teaspoons) and urine will be collected for routine tests.
* You may also have a CT scan and/or MRI to check the status of the disease.

Long-Term Follow-Up:

After the end-of-study visit, you will have a study visit every month for the first year and then once a year for 10 years. At these visits, you will have a physical exam.

You may also have CT scans and/or MRIs every 8 weeks for the 1st 6 months, every 3 months for the next year, then every 6 months for 1 1/2 years, and then at least 1 time a year after that. This will be done to check the status of your disease.

Researchers would like to keep track of your medical condition and some general health information about you through yearly follow-up visits, letters, and/or phone contact, for up to 10 years. More information (such as other treatments and/or disease response) will be collected if follow-up studies show changes in the disease or in your overall health.

If the disease has gotten worse, researchers will keep track of which parts of your body are involved. Researchers will also collect information about any other cancers or major organ problems you might have developed. Keeping in touch with you and checking on your condition will help researchers look at the long-term effects of the study.

This is an investigational study. Doxercalciferol is FDA approved and commercially available for reducing high levels of a hormone in patients undergoing chronic renal dialysis. Its use in this study, for this disease, is investigational.

Up to 24 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntary consent obtained from the patient or their legal guardians.
2. Patient must be greater than 2 and less than 26 years old at time of study entry or at time of initial diagnosis
3. Patient must have had histologic verification of a solid malignancy at initial diagnosis (excluding brain stem tumors and visual pathway gliomas)
4. Patient must have recurrent measurable or evaluable disease after therapy or refractory to conventional therapy with presence of disease confirmed by standard imaging or biopsy
5. Must start protocol therapy within two weeks of disease evaluation and determination of eligibility.
6. Performance status of >20% on Lansky play scale for subjects <10 years of age, >20% on Karnofsky score for subjects >= 10 years of age
7. Patient must have fully recovered to less than or equal to grade 1 from the acute toxic effects of prior therapy, to meet eligibility criteria
8. Adequate bone marrow function defined as peripheral absolute neutrophil count (ANC) equal or more than 500/mm^3, Hemoglobin equal or more than 8g/dl, Platelets equal or more than 20,000/mm^3
9. Adequate renal function defined as serum creatinine <1.5 X upper limit of normal (ULN) or age adjusted creatinine clearance of >70ml/min/1.73m^2
10. Adequate liver function defined as total bilirubin <1.5 X upper limit of normal (ULN) and AST <2 X upper limit of normal (ULN)
11. Serum calcium, phosphorus, or PTH levels must be </= to the upper limit of normal age adjusted values per institutional guidelines.
12. Urine calcium level must be </= to the upper limit of normal value per institutional guidelines
13. Women of childbearing potential must have a negative serum or urine pregnancy test and not be breastfeeding prior to study therapy. Women of childbearing potential must be using an adequate form of contraception to avoid pregnancy during therapy and for at least 4 weeks after the end of study therapy in such a manner that the risk of pregnancy is minimized (Women of childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization)

Exclusion Criteria:

1. Any past history of urine calcium stones, idiopathic hypercalcemia, hereditary bone disease, or hypercalciuria in the subject
2. Concurrent Medications: Patients currently taking digitalis or thiazides are ineligible
3. Concurrent Medications: Oral calcium and vitamin D supplements and all homeopathic medications must be discontinued 2 weeks prior to study entry and while on study therapy.
4. Use of other anti-tumor therapy, including but not limited to chemotherapy, radiation therapy, immunotherapy, other investigational agents or other biologic therapy, during study therapy, with the exception of palliative radiation therapy to non-index lesions.

Ages: 2 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continual reassessment method during 28 day cycles, weekly visits for first cycle and monthly for each additional cycle

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Zage, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org